CLINICAL TRIAL: NCT04743687
Title: The Efficacy and Safety of Zanuburutinib in Relapsed and Refractory Idiopathic Multicentric Castleman Disease (iMCD): a Prospective, Single-center, Single-arm Trial
Brief Title: Zanuburutinib in Relapsed and Refractory iMCD: a Prospective, Single-center, Single-arm Trial
Acronym: iMCD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZS-2551
Record Dates: First submitted 2021-02-03; First posted 2021-02-08 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Idiopathic Multicentric Castleman's Disease
Keywords: iMCD; Zanuburutinib; efficacy; safety
MeSH Terms: conditions — Multi-centric Castleman's Disease | interventions — zanubrutinib

STUDY DESIGN:
Intervention Model Description: This will be a single center, single arm, phase 2 study.
Masking Description: This will be an open label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Zanuburutinib (Experimental): Oral Zanuburutinib 160mg twice a day
  Interventions: Drug: Zanubrutinib

INTERVENTIONS:
Drug: Zanubrutinib — Oral Zanuburutinib, 160mg twice a day
  Other Names: brukinsa

SUMMARY:
To explore the effectiveness and safety of Zanuburutinib in relapsed and refractory idiopathic Multicentric Castleman's disease (iMCD) patients.

DETAILED DESCRIPTION:
This is a single center, open-labeled , single arm, prospective study which includes a safety run-in phase. The primary endpoint is the overall response rate which includes complete response (CR) and partial response (PR) at Week 12 and Week 24. The secondary endpoints include progression-free survival (PFS), overall survival (OS), and adverse events. There are two phases of the study. The first phase is the 'safety run-in phase'which plans to enroll 6 patients who would be observed for safety issues for 12 weeks after study drug administration. If no Grade ≥ 4 (CTCAE) adverse events (AE) occurs during this phase, the study would enter the second phase; if Grade ≥ 4 (CTCAE) AE happens during this phase, the study would be terminated. In the second phase of the study, another 24 patients would be enrolled. All enrolled patients would receive the study drug until progression of disease, intolerability of the drugs or Week 96 and would be followed every 4 weeks in the first 12 weeks, every 12 weeks until Week 48 and every 24 weeks until Week 96. The follow-up phase to assess PFS and OS will last from initiation of study drug to 36 months after enrollment (evaluation would be carried out every 24 weeks after Week 96). The total study duration will be 4 years after the last patient starts study medication.

ELIGIBILITY:
Inclusion Criteria:

* fulfilled the CDCN (Castleman Disease Collaborative Network) diagnostic criteria of iMCD
* relapsed or refractory disease. Relapsed = patients who ever achieved overall partial response (PR) or complete response (CR) with prior lines of therapy suffered from progressive disease (PD); refractory = iMCD patients who never achieved PR or CR with the first-line treatment but suffered from PD during treatment.
* Eastern Cooperative Oncology Group performance status (ECOG-PS ≤ 2)
* Neutrophil count ≥ 0.75×10^9/L, hemoglobin ≥ 70 g/L and platelet count > 30×10^9/L
* Total bilirubin ≤ 2 x ULN (upper limit of normal), AST（aspartate aminotransferase） or ALT（Alanine aminotransferase）≤ 2.5 x ULN
* INR （international normalized ratio) and APTT(activated partial thromboplastin time) ≤ 1.5 x ULN；eGFR>25ml/min/1.73m2
* estimated survival ≥ 3 months
* agree to take birth control methods during study period for women of reproductive age
* agree to provide informed consent

Exclusion Criteria:

* concurrent malignancies
* prior history of receiving any kind of BTK (Bruton's tyrosine kinase) inhibitors
* patients with SLE (systemic lupus erythematosus), HHV-8 (human herpesvirus-8) infection or POEMS syndrome
* History of major surgery or radiation therapy within 4 weeks before initiation of study drug
* history of myocardial infarction within 1 years
* patient with history of heart failure (NYHA 3 or 4) would be excluded unless his LVEF(left ventricular ejection fraction) ≥ 50% within 1 months
* primary cardiomyopathy; Qtc > 450ms for men and > 470ms for women
* breast feeding or pregnant women
* intolerance for oral regimen due to gastro-intestinal disorders
* uncontrolled infection
* positive HBV(hepatitis B virus)-DNA titers or positive HbsAg; positive HCV(hepatitis C virus)antibody; patients with HIV infection
* patients with history of bleeding disorders
* cerebral infarction or intracranial bleeding within 6 months
* active bleeding disorders within 2 months
* taking anti-platelet or anticoagulation drugs
* taking drugs which strongly inhibit P450 CYP3A
* patients or their relatives fail to understand the purpose of the study
* any other conditions that the investigators consider to be not appropriate for inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) at Week 12 | From date of treatment initiation to 12 weeks after treatment
  Overall response (including partial response and complete response) rate at week 12 after zanuburutinib therapy
Overall response rate (ORR) at Week 24 | From date of treatment initiation to 24 weeks after treatment
  Overall response (including partial response and complete response) rate at week 24 after zanuburutinib therapy

SECONDARY OUTCOMES:
Progression free survival | From date of treatment initiation until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  Time to disease progression or death
Overall survival | From date of treatment initiation until the date of death from any cause, whichever came first, assessed up to 36 months
  Time to death
Number of Participants With Treatment-related Adverse Events | From initiation study regimen to 3 months after the end of treatment or to time point of the initiation of second line therapy
  Number of Participants With Treatment-related Adverse Events as Assessed by CTCAE v4.0 ( ≥1 Grade)

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang L, Gao YH, Li SY, Zhao H, Zhang MY, Yu YY, Liu YT, Li J. A prospective study of zanubrutinib, a Bruton tyrosine kinase inhibitor, in relapsed/refractory idiopathic multicentric Castleman disease. Int J Hematol. 2024 Jun;119(6):631-637. doi: 10.1007/s12185-024-03747-7. Epub 2024 Mar 28. PMID 38546960